CLINICAL TRIAL: NCT03325842
Title: Transcultural Validation of Activities Scale for Kids (ASK):Estimate of the Reliability of the Italian Version in the Population With PCI
Brief Title: Transcultural Validation of Activities Scale for Kids (ASK)
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Stefania Costi, Researcher in PT, University of Modena and Reggio Emilia
Other Study IDs: ASKp_PCI_UDGEE
Record Dates: First submitted 2017-10-24; First posted 2017-10-30 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy and Healthy Individuals
Keywords: Cross-cultural comparison; Disability evaluation; Self-assessment; Child; Adolescent
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral palsy: ASKp will be submitted to children of 5 to 15 years with hemiplegia or diplegia due to Cerebral Palsy, with normal or slightly impaired cognitive level.
  Interventions: Diagnostic Test: ASKp
- Healthy individuals: ASKp will be submitted to children of 5 to 15 years with typical development
  Interventions: Diagnostic Test: ASKp

INTERVENTIONS:
Diagnostic Test: ASKp — 30 items questionnaire

SUMMARY:
The Activities Scale for Kids performance (ASKp) is one of the few self-assessment questionnaires in pediatric rehabilitation that measures child perception in performance of daily routine activities. ASKp is composed of 30 questions designed to explore activities and participation in children and teenagers with musculoskeletal disorders. Scores assess level of physical ability, identify appropriate treatment and monitor changes over time. We recently undertook the cross-cultural validation to achieve a culturally adapted Italian version of ASKp: the Italian version is now to be tested on Italian children.

DETAILED DESCRIPTION:
The purpose of the study isto test the psychometric properties of the Italian version of the ASKp assessment scale, in a representative sample of individuals with PCI.

ASK p will be administered on a sample of individuals belonging to the population of children and / or adolescents with diplegia and hemiplegia as a consequence of PCI. We will perform comprehensive descriptive analysis of the data collected as well as the measurement of the degree of reliability of the Italian version of the scale. The aim is to obtain an estimate of ASKp reliability obtained through transcultural validation.

Additionally, we will submit the ASKp on a control group of typical development children in order to test its ability to discriminate between different skill levels.

ELIGIBILITY:
Inclusion Criteria:

* Italian nationality

Exclusion Criteria:

* moderate or severe cognitive impairment;
* linguistic barriers

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children or adolescents and children or adolescents with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Split-half reliability analysis by alpha of Cronbach, one item out. | 1 day
  A split-half reliability analysis will be performed by calculating the alpha of Cronbach by removing one item at a time. It will then be assessed which items lower the degree of internal reliability of the questionnaire. Items that reduce internal consistency will be eliminated and the final alpha will be calculated. For a group of children with PCI and for the control group a comprehensive descriptive analysis of the collected data will be performed, representing the distribution of scores obtained by age group.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Ferrari, MD, Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Arcispedale Santa Maria Nuova, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fabbri L, Neviani R, Festini F, Costi S. Transcultural validation of Activities Scale for Kids (ASK): translation and pilot test. Acta Biomed. 2016 May 26;87 Suppl 2:70-9. PMID 27240035
- [Derived] Costi S, Filippi MC, Braglia L, Beccani L, Corradi I, Bruzzi E, Signorelli C, Pelosin E. Reliability and construct validity of the Activities Scale for Kids in Italian children with cerebral palsy. Disabil Rehabil. 2022 Oct;44(21):6445-6451. doi: 10.1080/09638288.2021.1966519. Epub 2021 Aug 20. PMID 34415225
- [Derived] Costi S, Mecugni D, Beccani L, Alboresi S, Bressi B, Paltrinieri S, Ferrari A, Pelosin E. Construct Validity of the Activities Scale for Kids Performance in Children with Cerebral Palsy: Brief Report. Dev Neurorehabil. 2020 Oct;23(7):474-477. doi: 10.1080/17518423.2020.1764649. Epub 2020 Jun 7. PMID 32508188